CLINICAL TRIAL: NCT04691453
Title: Randomized Clinical Trial Comparing the Oncology Outcome and Safety of QM-B and QM-C Hysterectomy for Early Cervical Cancer
Brief Title: QM-B and QM-C Hysterectomy for Early Cervical Cancer
Acronym: QMBCHECC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southern Medical University, China (Other)
Responsible Party: Principal Investigator, Chen Chunlin, Director, Head of Obstetrics and Gynecology, Principal Investigator, Clinical Professor, Southern Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2020-175
Record Dates: First submitted 2020-10-20; First posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Uterine Cervical Neoplasms
Keywords: Cervical cancer; QM-B; QM-C; Oncology outcome; Safety; Hysterectomy; Radical Hysterectomy; Abdominal
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QM-C Hysterectomy (Active Comparator): QM-C Hysterectomy
  Interventions: Procedure: QM-C Hysterectomy
- QM-B Hysterectomy (Experimental): QM-B Hysterectomy
  Interventions: Procedure: QM-B Hysterectomy

INTERVENTIONS:
Procedure: QM-C Hysterectomy — This operation corresponds to the classical radical hysterectomy. The lateral border is defined as the medial aspect of the internal iliac artery and vein. Transection of the rectovaginal and rectouterine ligaments is performed at the rectum. Transection of the ventral parametrium ligament is performed at the bladder. Both the vesicouterine and vesicovaginal ligaments are resected. The ureter is completely mobilized and lateralized. The length of the vaginal cuff is adjusted to the vaginal extent of the tumor.
  Other Names: Type III radical hysterectomy; Radical hysterectomy; Type C radical hysterectomy
  Arms: QM-C Hysterectomy
Procedure: QM-B Hysterectomy — Type B is the modified radical hysterectomy. The ureter is unroofed and mobilized laterally, permitting transection of the paracervix at the level of the ureteral tunnel. Partial resection of the uterosacral peritoneal fold of the rectouterine ligament (dorsal parametrium) and the vesicouterine (ventral parametrium) ligament also is a standard component of this resection. Approximately 10 mm of the vagina from the caudal edge of the cervix or tumor is resected, without intent to radically resect the paravaginal tissues.
  Other Names: Type II radical hysterectomy; Modified radical hysterectomy; Type B radical hysterectomy
  Arms: QM-B Hysterectomy

SUMMARY:
The goal of this clinical research study is to compare the long-term outcomes and safety of Querleu-Morrow-B(QM-B) and Querleu-Morrow-C(QM-C) hysterectomy for early cervical cancer. In this study, the surgical approach for QM-B and QM-C hysterectomy will be abdominal.

DETAILED DESCRIPTION:
Primary Objective:

To compare 5-year overall survival and 5-year disease-free survival amongst patients who undergo a QM-B hysterectomy versus those who undergo a QM-C hysterectomy for early stage cervical cancer.

Secondary Objectives:

Compare operation time between arms. Compare blood loss between arms. Compare blood transfusion between arms. Compare intraoperative complications between arms. Compare postoperative complications between arms. Compare quality of lifes between arms.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have signed an approved Informed Consent
* 18.5≤BMI<28
* Histologically confirmed primary adenocarcinoma, squamous cell carcinoma or adenosquamous carcinoma of the uterine cervix;
* Patients with Histologically confirmed stage IA1 (with lymph vascular invasion), stage IA2, stage IB1, stage IB2, or stage IIA1 disease(FIGO 2018).
* Eastern Cooperative Oncology Group(ECOG) Performance Status of 0 or 1.
* Patients undergoing the Non-Fertility-Sparing surgery.
* Patients undergoing abdominal surgery.

Exclusion Criteria:

* The life expectancy of the patient is less than 6 months.
* Patients with serious medical diseases.
* Patients with contraindications to surgery or anesthesia.
* Preoperative imaging studies suggest metastasis to pelvic lymph nodes or para-aortic lymph nodes.
* Patient asks to preserve fertility.
* The patient requested direct radiation therapy.
* Patients with adjuvant radiotherapy or chemotherapy before surgery.
* Patients judged by the investigator to be unsuitable to participate in this trial.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 538 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Rate of overall survival | 5 years from surgery
  Compare treatment equivalence
Rate of disease-free survival | 5 years from surgery
  Compare treatment equivalence

SECONDARY OUTCOMES:
Operation time | Intra-operatively
  Compare operation time between groups by timer
Volume of blood loss | Intra-operatively
  Compare blood loss between groups by assessment
Rate of blood transfusion | Intra-operatively
  Compare rate of blood transfusion between groups
Rate of intraoperative complications | Intra-operatively
  Compare intraoperative complications between groups
Rate of postoperative complications | 6 months from surgery
  Compare postoperative complications between groups
Quality of life Questionnaires | 6 months from surgery
  Compare quality of lifes between groups by questionnaire: EORTC CX24. EORTC CX24 for symptom experience, body imageand sexual/vaginal functioning. The scores of EORTC CX24 range from 0 to 100; a higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms.
Pelvic Floor Distress Inventory Questionnaire | 5 years from surgery
  Compare PFDI between groups by questionnaire PFDI-20. The calculation of the total scores of PFDI-20 range from 0 to 300; the higher the score the greater the perceived impact that pelvic floor dysfuntion has on a patient's life.
Costs | 6 months from surgery
  Compare costs between groups

CONTACTS AND LOCATIONS:
Overall Officials: Chunlin Chen, Doctor, Study Chair — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Obstetrics and Gynecology, Nanfang Hospital, Southern Medical University, No. 1838, Guangzhou Avenue, Guangzhou 510515, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No